CLINICAL TRIAL: NCT02270723
Title: Effect of Colloid Versus Crystalloid on Coagulation in Elective Urological Surgery
Brief Title: The Effect of Human Albumin on Coagulation Competence and Hemorrhage
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Kirsten Cleemann Rasmussen (Other)
Responsible Party: Sponsor-Investigator, Kirsten Cleemann Rasmussen, MD, Specialist in Surgery, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COL18
Record Dates: First submitted 2014-09-27; First posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Hemorrhage; Complicating Delivery, Coagulation Defect
MeSH Terms: conditions — Hemorrhage; Hemostatic Disorders | interventions — Serum Albumin, Human; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Human Albumin " Behring" (Active Comparator): Infusion of 5% Human Albumine, maximal 25 ml/kg, is administered intravenously during anaesthesia, duration up to 6 hours
  Interventions: Drug: 5% Human Albumin " Behring"
- Lactated Ringer (Placebo Comparator): Infusion of Lactated Ringer solution 25 ml/kg, is administered intravenously during anaesthesia, duration up to 6 hours
  Interventions: Drug: Lactated Ringer

INTERVENTIONS:
Drug: 5% Human Albumin " Behring" — Intravenous infusion of 5% Human Albumin during major surgery
  Other Names: Human Albumin
  Arms: Human Albumin " Behring"
Drug: Lactated Ringer — Intravenous infusion of Lactated Ringer during major surgery
  Other Names: Ringer
  Arms: Lactated Ringer

SUMMARY:
In a randomized clinical trial, the purpose is to investigate if perioperative coagulation and hemorrhage is influenced by colloid or crystalloid.

DETAILED DESCRIPTION:
5% Human Albumin is used for fluid therapy during surgery. This study evaluate whether affected coagulation competence induced by Human Albumin leads to a significant perioperative blood loss when compared to administration of lactated Ringer´s solution.

Data are gathered by the investigators, analysed by the sponsor, and remain confidential throughout the process. The investigators shall be involved in all stages of the study development and vouch for the completeness and accuracy of the data. No third part shall influence the protocol, trial conduct, data analysis, or reporting.

The investigators will include 40 patients undergoing cystectomy. Heart rate, mean arterial pressure, cardiac output are measured after induction of anaesthesia and insertion of the arterial catheter (T0), after establishing normovolaemia but before surgery (T1), after resection of the urinary bladder (T2), at the end of the surgery (T3), and two hours thereafter in the recovery room (T4).

Arterial blood is drawn for whole blood viscoelastic haemostatic assays to record clot initiation (R-Time), formation (Maximal Amplitude, MA), alpha angle(α) and lysis (Ly30) depicting haemostatic competence (thrombelastography). The investigators analyze blood for haemoglobin, creatinine, platelets, and fibrinogen. Furthermore, blood is drawn from the central venous catheter for lactate and blood gas variables (ABL 825, Radiometer, Copenhagen, Denmark). To avoid excessive administration of Human Albumin, patients receive lactated Ringer´s solution if considered needed after the infusion 25 mL/kg of the allocated fluid (non-study fluid).

The fluid balance inclusive the blood loss was calculated after cystectomy, at the end of surgery, and two hours thereafter. The investigators register complications postoperatively inclusive hospital stay until discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patient more than 18 years old
* Indication for elective post-renal operation including cystectomy
* Patient without anticoagulative, acetylsalicylic acid or nonsteroidal antiinflammatory drug

treatment for the last 5 days

Exclusion Criteria:

* Intracerebral bleeding, manifest cardiac insufficient, renal insufficient demanding dialysis, hepatic or coagulation diseases
* Pregnant or nursing
* Allergic to Human Albumin
* Disturbance in electrolytes
* Patient under committee
* Patient joining another trial interfering the actual trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-08 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Measurement of coagulation during surgery and in the recovery room | up to 1 day after surgery
  Changes in fibrinogen, platelets, hemoglobin, alpha angle and maximum amplitude

SECONDARY OUTCOMES:
Measurement of postoperative surgical complications | From date of operation up to 1 months postoperatvely
  Numbers of participants with site infection, postoperative bleeding and leak requiring reoperation
Measurement of hemorrhage and use of blood products during anesthesia and in the recovery room | up to 1 day after surgery
  Volume of lost blood during anesthesia, infusion of blood products, lactated Ringer's and Human Albumin

CONTACTS AND LOCATIONS:
Overall Officials: Niels H Secher, MD PHD Prof, Study Chair — Rigshospitalet, University of Copenhagen
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Rasmussen KC, Hojskov M, Johansson PI, Kridina I, Kistorp T, Salling L, Nielsen HB, Ruhnau B, Pedersen T, Secher NH. Impact of Albumin on Coagulation Competence and Hemorrhage During Major Surgery: A Randomized Controlled Trial. Medicine (Baltimore). 2016 Mar;95(9):e2720. doi: 10.1097/MD.0000000000002720. PMID 26945358